CLINICAL TRIAL: NCT02314026
Title: Clinical Study of the BreathID® System to Train the Algorithm for the ¹³C-Octanoate Breath Test With or Without the ¹³C-Methacetin Breath Test (OBT and MBT Respectively) for Correlation With Histological Findings Associated With Non-Alcoholic Steatohepatitis (NASH) and Other Liver Diseases
Brief Title: BREATHID Octanoate Breath Test With or Without Methacetin Breath Test for Correlation With Biopsy in NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NASH-EX-1114
Record Dates: First submitted 2014-12-04; First posted 2014-12-10 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2019-02

CONDITIONS: Non-Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Suspected NASH (Experimental): 13C-Octanoate, 13C-Methacetin
  Interventions: Device: Suspected NASH BreathID test with 13C-Octanoate; Device: Suspected NASH Breath test with 13C Methacetin

INTERVENTIONS:
Device: Suspected NASH BreathID test with 13C-Octanoate — Subject will have breath measured before and after ingestion of solution of 100 mg 13C Octanoate dissolved in 150 cc of water
  Other Names: Sodium Octanoate breath test
Device: Suspected NASH Breath test with 13C Methacetin — Subject will have breath measured before and after ingestion of solution of 75 mg 13C Methacetin dissolved in 150 cc of water

SUMMARY:
This study's aim is to develop an algorithm for the ¹³C-Octanoate Breath Test with or without the ¹³C-Methacetin Breath Test (OBT and MBT respectively) for correlation with histological findings associated with of Non-Alcoholic Steatohepatitis (NASH) and other liver diseases using the BreathID® System

DETAILED DESCRIPTION:
Non-Alcoholic Steatohepatitis (NASH) is a growing epidemic in the western world due to the contemporary eating habits and life styles.NASH can lead to cirrhosis, hepatic carcinoma and other liver complications. There are currently some treatments available. The only definitive way of detecting NASH in patients with advanced liver disease is by liver biopsy. However, liver biopsy has disadvantages, such as sampling errors, chance of complications and does not lend itself to following up after treatment.

A non-invasive test that could potentially replace biopsy and aid in NASH detection and treatment monitoring, would improve management of suspected NASH patients without the need for biopsy. This protocol will obtain the results of one or two different breath tests to provide an accurate evaluation of the liver status in patients at high risk for NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women (≥18 years of age)
2. Liver biopsy, indicating NAFLD/NASH, performed within 6 months prior to both breath tests OR undergoing liver biopsy to rule-out or confrim NAFLD/NASH. NOTE:The samples obtained meet defined quality criteria. (In Appendix II of protocol)
3. Any elevation of liver enzymes above the upper limit of normal (any or all of the following: AST, ALT, GGT, Alkaline phosphatase) for at least 3 months
4. No other known co-existent liver disease, excluded by appropriate serologic / other testing
5. Imaging - US / CT / MRI (if available) with the typical image of Fatty Liver or suggestive of NASH.
6. Patient (or legal guardian) able and willing to sign an Informed Consent Form
7. Can tolerate an overnight (8-hour) fast

Exclusion Criteria:

1. Positive studies for any of the following within three years prior to biopsy:

   1. Anti HCV positive
   2. Anti HB core antibody positive
   3. Iron saturation > 60% + gene test for hereditary hemochromatosis or iron overload as defined by presence of 3+ or 4+ stainable iron on liver biopsy
   4. Antinuclear antibody at a titer > 1: 160 along with hypergammaglobulinemia and 5 times ALT normal levels
   5. Alpha-1-antitrypsin level below lower limit of normal (< 150 mg/dl) or no PAS diastase resistant globules on biopsy.
   6. Primary biliary cirrhosis as defined by elevation of alkaline phosphatase greater than upper limit of normal and anti-mitochondrial antibody (AMA) of greater than 1:80 and consistent liver histology
   7. Low level of ceruloplasmin
   8. Drug-induced liver disease as defined on the basis of typical exposure and history
2. Patients known to have chronic liver disease other than NAFLD as routinely diagnosed by the investigator
3. Concurrent acute hepatic condition other than NAFLD
4. Alcohol consumption > 20 gm/day (0.71 oz/day) for women and > 30 gm/day (1.06 oz/day) for men
5. Drugs that may interfere with octanoate metabolism or can also cause NAFLD independent of the metabolic syndrome, including: corticosteroids, amiodarone, tetracycline, valproic acid, methotrexate, stavudine, zidovudine
6. When MBT is performed subject should not have taken any of the following at least 48 hours prior to the breath test: Acyclovir , allopurinol, carbamazepine, cimetidine, ciprofloxacin, daidzein, (herbal) disulfiram, echinacea, enoxacin, famotidine, fluvoxamine, methoxsalen, mexiletine, montelukast, norfloxacin, phenylpropanolamine, phenytoin, propafenone, rifampin, terbinafine, ticlopidine, thiabendazole, verapamil, zileuton or any medication that might interfere with Methacetin metabolism or might affect CYP 1A2
7. Patients that have had more than 10% weight change between biopsy and enrollment.
8. Hypersensitivity to any of the study substrates; i.e. Octanoate or Methacetin respectively
9. Known extra-hepatic diseases including but not limited to: severe congestive heart failure (NIHA>2), known severe pulmonary hypertension (>35 mmHg), history of chronic obstructive pulmonary disease or uncontrolled symptomatic bronchial asthma or uncontrolled diabetes mellitus (HA1c>9.5%)
10. Previous surgical GI bypass surgery
11. Extensive small bowel resection (>100 cm)
12. Known uncontrolled malabsorption or diarrhea
13. Concurrent total parenteral nutrition
14. Any organ transplant
15. Patients receiving any anti-viral treatment or any other liver directed therapy, procedure or surgery between the time of the biopsy and the breath test
16. Pregnant or breast feeding
17. Patients and/or legal guardian unable or refusing to sign informed consent
18. Patients that, based on the opinion of the investigator, should not be enrolled into this study due to safety / adherence reasons.
19. Patients participating in other clinical trials and already receiving experimental treatments or procedures
20. Patients with suspected or documented hepatocellular carcinoma by ultra-sound or other imaging modality
21. Patients diagnosed with partial / complete portal venous occlusion, hepatic venous occlusion, previous PHT surgery, or placement of a transjugular intrahepatic portosystemic shunt (TIPS) according to initial imaging studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, M.D., Study Director — Hadassah Medical Organization
Locations (11):
- United States (8):
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - San Antonio Military Medical Center, Forts Sam Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Liver Associates, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Mary Immaculate Hospital, Newport News, Virginia
  - St. Mary's Hospital, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Antwerp University Hospital (UZA), Edegem, Belgium
- Hôpital Pitié Salpêtrière, Paris, France
- Freeman Hospital, Newcastle, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suspected NASH
Started | 135
Completed | 107
Not Completed | 28
Not completed — Protocol Violation | 28

BASELINE CHARACTERISTICS:
Arm/Group | Suspected NASH
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 15
  United States | 102
  United Kingdom | 9
  France | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy Proven Non-Alcoholic Steatohepatitis
Description: Non-Alcoholic Steatohepatitis (NASH) as determined by liver biopsy histology will be the comparator
Time Frame: 30 days
Population: Subjects that had a valid biopsy and performed both Octanoate and Methacetin Breath test
Measure: Count of Participants; unit: Participants
Arm/Group | Suspected NASH
Number analyzed (Participants) | 107
Participants
  Definite NASH | 74
  Probable NASH | 20
  Absent of NASH | 13

2. Primary Outcome: Liver Decompensation as Measured by Area Under Receiver Operating Curve
Description: Observe if breath tests correlate to clinical outcome of liver decompensation, including ascites, variceal bleeding, hepatic encephalopathy and spontaneous bacterial peritonitis.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Suspected NASH
Number analyzed (Participants) | 107
Probability | 0.852 [0.771 to 0.933]

3. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: A phone call will be made to each subject 48 hours after the last breath test to confirm that no adverse events related to breath test have been experienced.
Time Frame: 48 hours from last breath test
Measure: Count of Participants; unit: Participants
Arm/Group | Suspected NASH
Number analyzed (Participants) | 135
Participants
  Possibly related adverse event | 0
  No possibly related reported adverse events | 135

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 36 months from enrollment
Arm/Group | Suspected NASH
All-Cause Mortality (participants affected / at risk) | 0/135
Serious Adverse Events (participants affected / at risk) | 1/135
Other Adverse Events (participants affected / at risk) | 5/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suspected NASH (N=135)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) — Acute cholecystitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suspected NASH (N=135)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Patient suffered from abdominal pain and cramping
Nausea (Gastrointestinal disorders) | 2 (2) — Patient suffered from nausea on day of test
Dizziness (Nervous system disorders) | 1 (1) — Patient suffered from dizziness
Headache (Nervous system disorders) | 1 (1) — Patient suffered from headache on day of test

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT02314026/Prot_SAP_000.pdf